CLINICAL TRIAL: NCT01005927
Title: Fructooligosaccharide and Calcium Absorption in Adolescent Girls
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Abbott Nutrition (Industry); GTC Nutrition (Industry)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GTC Study
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: Calcium; Bone and Bones; Girls; Bone Mineralization; Fiber; Fructooligosaccharide; Female; Healthy; Adolescents
MeSH Terms: conditions — Osteoporosis | interventions — fructooligosaccharide; Dietary Fiber; Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Fructooligosaccharide (Placebo Comparator): 0 g fructooligosaccharide added to calcium-containing beverage
  Interventions: Dietary Supplement: Fructooligosaccharide
- 3 g Fructooligosaccharide (Active Comparator): 3 g fructooligosaccharide added to calcium-containing beverage
  Interventions: Dietary Supplement: Fructooligosaccharide

INTERVENTIONS:
Dietary Supplement: Fructooligosaccharide — Zero or 3 g of a fructooligosaccharide will be administered in a beverage containing 300 mg total calcium as well as 15 mg 44Ca (calcium carbonate). Participants will be given one of the above beverages in addition to intravenously receiving 5 mg 43Ca (calcium chloride)in 10 ml saline.
  Other Names: Fiber and Calcium

SUMMARY:
Fructooligosaccharides (FOS) are believed to have positive effects on calcium absorption and bone accrual during growth. This study aims to see whether the addition of fiber in the form of FOS to a calcium-containing beverage will increase calcium absorption. During two clinical visits, participants will receive a beverage containing a small amount of calcium, supplemented with either no dietary fiber or a small amount of fiber. Height, weight, bone density and geometry, calcium absorption, and physical fitness will be measured. The effects of this fiber intervention may provide support for improving bone health with minimal fiber supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Calcium intake of 900-1300 mg/d
* Generally healthy

Exclusion Criteria:

* Male
* BMI > 90th percentile for age
* Takes medication that influences calcium metabolism
* Any disorder of calcium or bone homeostasis (hypercalcemia, Paget's Disease)
* Smoking, illegal drug consumption
* Any gastrointestinal disease (Crohn's Disease, Celiac Disease, Inflammatory Bowel Disease)

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Fractional Calcium Absorption | 24 h urine and 3 h blood

SECONDARY OUTCOMES:
Bone density and geometry measured with peripheral quantitative computed tomography (pQCT) | Initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Purdue University; Berdine R Martin, PhD, Study Director — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States